CLINICAL TRIAL: NCT00472342
Title: The Effects of Exercise on Adipokine in Impaired Fasting Glucose or Impaired Glucose Tolerance Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: kenshin46
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2007-05-11 (Estimated); Status verified 2007-05

CONDITIONS: Impaired Glucose Tolerance; Diabetes
Keywords: impaired glucose tolerance; impaired fasting glucose; diabetes; adipokine; adiponectin; RBP-4; adrenomedullin
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: exercise prescription

SUMMARY:
Many adipokines are thought that related with metabolic disturbance such as glucose intolerance, dyslipidemia, and insulin resistance. It is reported that regular physical training could prevent the progression of diabetes from prediabetes and improve the insulin resistance. After physical training, many adipokine levels were changed due to improving insulin resistance.

In this study, we will examine the various adipokine levels such as adiponectin, RBP-4, and adrenomedullin after exercise training through exercise prescription in IFG and IGT patients.

DETAILED DESCRIPTION:
Backgrounds: Type 2 diabetes mellitus can be caused by genetic and environmental factors. Type 2 diabetes could be prevented by modifying the environmental risk factors such as physical inactivity, heavy eating, and obesity. It is reported that regular physical training could prevent the progression of diabetes from prediabetes such as impaired glucose tolerance (IGT) and impaired fasting glucose (IFG).

Prediabetes, the term of IGT and IFG, could progress to type 2 diabetes in 30~40 % within 4~5 years. Moreover, cardiovascular and cerebrovascular events are increased in prediabetic patients like as type 2 diabetic patients.

Adipose tissue is thought as a endocrine organ that secrets and regulates various hormones known as adipokines including adiponectin, resistin, leptin, visfatin, tumor necrosis factor (TNF)-α, interleukin-6 (IL-6), and retinol-binding protein 4 (RBP 4). Recently, many adipokines are thought that related with metabolic disturbance such as glucose intolerance, dyslipidemia, and insulin resistance.

Adiponectin is known as anti-diabetic factor exerting actions on muscle fatty acid oxidation and insulin sensitivity. Plasma adiponectin levels are significantly decreased in obese, type 2 diabetes, and insulin resistant patients and correlated with insulin sensitivity. Also, adiponectin has anti-inflammatory and anti-atherogenic effects. So, adiponectin is representative insulin sensitivity marker and may be a protective factor against development of type diabetes. In previous data, there was discrepancy in effects of exercise on adiponectin levels. Some study showed exercise interventions could not have effects on adiponectin levels. However, other study suggested that physical fitness may increase adiponectin levels in obese insulin resistant adults.

RBP-4, secreted by adiocytes, has effects on reducing glucose transporter 4 (GLUT 4) in adipocytes or increasing gluconeogenesis enzyme activity such as PEPCK in the liver. Also, it is known that RBP-4 is elevated in insulin resistant patients such as type 2 diabetes and obesity. After exercise training, RBP-4 levels were decreased in subjects with improvements of insulin resistance.

Adrenomedullin (AM), originally isolated in pheochromocytoma, is recently reported as adipokine. AM is highly expressed in adipocyte of high fat diet mice or obese rat model and elevated in type 2 diabetic patients. Also, AM expression on white and brown adipose tissue was increased after adrenergic stimulation. So, it is expected that AM expression will be changed by exercise.

In this study, we will examine the various adipokine levels such as adiponectin, RBP-4, and adrenomedullin after exercise training through exercise prescription in IFG and IGT patients.

Methods

Subjects Subjects having IFG and IGT on the basis of a 75g oral glucose tolerance test (OGTT) according to American Diabetes Association criteria will be studied.

Inclusion Criteria

1. Age; 30~70
2. Subjects with IGT and IFG
3. Subjects with having possibility of exercise stress test
4. Subjects with having a strong will to this study

Exclusion Criteria

1. Age <30 or >70
2. Cr more than 1.5 mg/dL
3. AST, ALT levels more than twice as upper normal range
4. Subjects having past history of coronary artery disease

Study design

1. Study design - before and after methods
2. Visit time - baseline, after 3months, after 6months
3. 1st visit- IGT and IFG diagnosis by 75g OGTT fill up the agreement Lab sampling
4. 2nd visit - exercise stress test exercise prescription by physician follow wup lab sampling
5. 3rd visit - follow up lab sampling completing the study
6. Dietary pattern data - FFQ and 3 day dietary recall Baseline - FFQ and 3 day dietary recall 2nd visit - 3 day dietary recall 3rd visit - 3 day dietary recall After 1 year - FFQ
7. Exercise pattern data - International Physical Activity Questionnaire (IPAQ)

1st, 2nd, and 3rd visits- IPAQ 8) We will compare the parameters according to results of IPAQ (by tertile) 9) We will adjust the parameters by dietary pattern 10) Anthropometric measurements

* Height, weight, BMI, waist circumference, hip circumference 11) Exercise capacity - exercise tolerance test and Vmax O2 12) Biochemical markers
* Glucose, HbA1C, WBC, AST, ALT, GGT, total cholesterol, triglyceride, HDL cholesterol, insulin, C-peptide 13) Adipokine
* adiponectine, RBP-4, adrenomedullin 14) Insulin resistance marker
* HOMA-IR 15) Inflammatory marker
* C-reactive protein (CRP)

ELIGIBILITY:
Inclusion Criteria:

1. Age; 30~70
2. Subjects with IGT and IFG
3. Subjects with having possibility of exercise stress test
4. Subjects with having a strong will to this study

Exclusion Criteria:

1. Age <30 or >70
2. Cr more than 1.5 mg/dL
3. AST, ALT levels more than twice as upper normal range
4. Subjects having past history of coronary artery disease

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2007-03; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Improvements of adipokine levels | 6 Months

SECONDARY OUTCOMES:
Prevention of diabetes | 1~5 year

CONTACTS AND LOCATIONS:
Overall Officials: Mi Young Lee, Dr, Principal Investigator — Department of Internal Medicine, Yonsei University Wonju College of Medicine; Choon Hee Chung, professor, Study Chair — Department of Internal Medicine, Yonsei Univerisity Wonju College of Medicine
Locations (1):
- Mi Young Lee, Wŏnju, Gangwon-do, South Korea